CLINICAL TRIAL: NCT01223092
Title: Genes and Gene Polymorphisms Associated With Infertility: Utilization of DNA Characteristics to Better Understand Reproductive Competence
Brief Title: Study of Gene Associations and Infertility
Status: Enrolling by invitation | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-00-10
Record Dates: First submitted 2010-10-08; First posted 2010-10-18 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Infertility
Keywords: IVF; infertility; DNA
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood serum, follicular fluid and sperm
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undegoing infertility treatment: Male and female patients undergoing infertility treatment

SUMMARY:
The purpose of this this study is to use DNA screening strategies to identify genes and localize genomic regions that are differentially expressed in patients with infertility to further understand the genetic basis for reproductive competence.

DETAILED DESCRIPTION:
Experimental strategies seek to discover small variants in DNA sequences, which are associated with certain infertility parameters. The alleles being analyzed in in vitro fertilization (IVF) population are sought to be associated with functional differences in the expression of the gene product that are then mechanistically linked to infertility.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing fertility care

Exclusion Criteria:

* none

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients undergoing infertility treamtnet
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2006-02; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of retrieved oocytes | 1 month

SECONDARY OUTCOMES:
Fertilization rate | 1 month
  Number of oocytes that are fertilized
Number of available embryos | 1 month
  Number of embryos that are available for transfer on day 3 or day 5
Pregnancy rates | 1 year
  Clinical pregnancy rates (detection of pregnancy hormone bHCG in blood) and delivery rates.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Franasiak, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

REFERENCES:
- [Background] Patounakis G, Treff N, Tao X, Lonczak A, Scott RT Jr, Frattarelli JL. The p53 codon 72 single nucleotide polymorphism lacks a significant effect on implantation rate in fresh in vitro fertilization cycles: an analysis of 1,056 patients. Fertil Steril. 2009 Oct;92(4):1290-1296. doi: 10.1016/j.fertnstert.2008.07.1783. Epub 2008 Oct 17. PMID 18930193
- [Derived] Patounakis G, Bergh E, Forman EJ, Tao X, Lonczak A, Franasiak JM, Treff N, Scott RT Jr. Multiple thrombophilic single nucleotide polymorphisms lack a significant effect on outcomes in fresh IVF cycles: an analysis of 1717 patients. J Assist Reprod Genet. 2016 Jan;33(1):67-73. doi: 10.1007/s10815-015-0606-z. Epub 2015 Nov 6. PMID 26545911